CLINICAL TRIAL: NCT05623228
Title: The Effectiveness and Efficacy of the Combination of the Integrated Psychological Therapy and Metacognitive Training in Schizophrenia and Treatment Resistant Schizophrenia. This is a Non-randomized Trial. The Therapy Lasts 60 Sessions.
Brief Title: The Effectiveness and Efficacy of the Combination of the Integrated Psychological Therapy and Metacognitive Training.
Acronym: ATHSCHIZ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rakitzi, Stavroula (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: (2022-2024); (ATH22-24) (Other: Dr. Stavroula Rakitzi private practice)
Record Dates: First submitted 2022-11-04; First posted 2022-11-21 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, treatment resistant schizophrenia, recovery
MeSH Terms: conditions — Schizophrenia; Schizophrenia, Treatment-Resistant | interventions — Drug Therapy; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Therapy Group A (Experimental): Therapy Group A Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  5 individuals with schizophrenia
  Interventions: Combination Product: The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia
- Therapy Group B (Experimental): Therapy Group B Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  2 individuals with schizophrenia
  Interventions: Combination Product: The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia
- Therapy Group C (Experimental): Therapy Group C Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  8
  Interventions: Combination Product: The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia
- Therapy Group D (Experimental): Therapy Group D Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  8
  Interventions: Combination Product: The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia
- Therapy Group E (Experimental): Therapy Group E Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  3
  Interventions: Combination Product: The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia
- Therapy Group F (Experimental): Therapy Group F Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  3
  Interventions: Combination Product: The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia
- Therapy Group G (Experimental): Therapy Group G Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented 3
  Interventions: Combination Product: The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia
- Therapy Group H (Experimental): Therapy Group H Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  3
  Interventions: Combination Product: The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia

INTERVENTIONS:
Combination Product: The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia — The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Other Names: Pharmacotherapy, rehabilitation

SUMMARY:
The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia.

Is it effective and efficacious?

DETAILED DESCRIPTION:
Individuals with schizophrenia and treatment resistant schizophrenia will participate on a group cognitive behavioral therapy and rehabilitation, in which Integrated Psychological Therapy and Metacognitive Training are going to be implemented. The therapy will last 60 biweekly sessions. This is a non randomized trial.

Speed of processing, working memory, verbal memory, visual memory, reasoning and problem solving, social cognition, symptoms, functional outcome and recovery will be evaluated before, after therapy and in a 6 months follow up.

MCCB, Social Perception Scale, the Greek Test for verbal memory, PANSS, WHO DAS 2. 0 (Greek), PSYRAT and the Recovery Assessment Scale will be used ih this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* No relapse and hospitalization
* Ambulant psychiatric treatment

Exclusion Criteria:

* Other psychotic disorders
* Relapse and hospitalization
* Substance abuse

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stavroula Rakitzi, Dr., Study Director — Private Practice
Locations (1):
- Stavroula Rakitzi, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Penney D, Sauve G, Mendelson D, Thibaudeau E, Moritz S, Lepage M. Immediate and Sustained Outcomes and Moderators Associated With Metacognitive Training for Psychosis: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2022 May 1;79(5):417-429. doi: 10.1001/jamapsychiatry.2022.0277. PMID 35320347
- [Background] Rakitzi, S., Georgila, P., Becker-Woitag, A.P. (2021). The recovery process for individuals with schizophrenia in the context of evidence based psychotherapy and rehabilitation. A systematic review. European Psychologist, 26(2), 96-111 doi/pdf/10.1027/1016-9040/a000400.
- [Background] Rakitzi S, Georgila P. Integrated Psychological Therapy and Treatment-Resistant Schizophrenia: Initial Findings. Psychiatry. 2019 Winter;82(4):354-367. doi: 10.1080/00332747.2019.1616658. Epub 2019 Aug 6. PMID 31385737
- [Result] Rakitzi S, Georgila P, Efthimiou K, Mueller DR. Efficacy and feasibility of the Integrated Psychological Therapy for outpatients with schizophrenia in Greece: Final results of a RCT. Psychiatry Res. 2016 Aug 30;242:137-143. doi: 10.1016/j.psychres.2016.05.039. Epub 2016 May 30. PMID 27280523
- [Result] Nuecterlein, K. H., & Green, M. F. (2006). MCCB. MATRICS Consensus Cognitive Battery. LA: MATRICS Assessment Inc.
- [Result] Fuentes, I., Garcia, S., Ruiz, J.C., Soler, J., & Roder, V. (2007). Social perception scale in Schizophrenia. A pilot study. International Journal of Psychology and Psychological therapy, 7 (1), 1-12.
- [Result] Kosmidou, M., & Vlahou, C. (2010). Greek verbal memory test. Athens: Parisianos.
- [Result] Lykouras, L., Botsis, A., & Oulis, P. (2005). Greek version of PANSS. Athens: Scientific publications.
- [Result] Haddock G, McCarron J, Tarrier N, Faragher EB. Scales to measure dimensions of hallucinations and delusions: the psychotic symptom rating scales (PSYRATS). Psychol Med. 1999 Jul;29(4):879-89. doi: 10.1017/s0033291799008661. PMID 10473315
- [Result] Hancock, N., Scanlan, J.N., Bundy, A.C., & Honey A. (2019). Recovery Assessment Scale -Domains & Stages (RAS-DS) Manual- Version 3. Sydney: University of Sydney.
- [Result] Koumpouros, Y., Papageorgiou, E., Sakellari, E. et al. (2018). Adaptation and psychometric properties' evaluation of the Greek version of WHODAS 2.0. Pilot application in Greek elderly population. Health Services and Outcomes Research Methodology,18(1), 63-74. https://doi.org/10.1007/s10742-017-0176-x.
- [Result] Aster, M., Neubauer, M., & Horn, R. (2006). Wechsler-Intelligenztest für Erwachsene WIE. Frankfurt: Harcourt Test Services
- See also: linkedin Stavroula Rakitzi — https://www.linkedin.com/
- See also: orcid: 0000-0002-5231-6619 — http://orcid.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: November 2022-Januar 2023 Patients were recruited from our private practice Dr. Stavroula Rakitzi Dr. Polyxeni Georgila
Pre-assignment Details: 35 patients with schizophrenia started
Groups:
- Therapy Group A: Therapy Group A Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  Monthly psychiatric treatment twice a week IPT and MCT, 60 minutes every session
  1. clozapine 350mg, amisulpride 200mg, mirtazapine 30 mg, clonazepam 2 mg
  2. olanzapine 22, 5 mg, alprazolami 0, 50 mg
  3. clozapine 200mg, 400 mg amisulpride, citalopram 20 mg, clonazepam 2 mg
  4. clozapine 300 mg, amisulpride 400mg
  5. 250mg clozapine, cariprazime 4, 5mg
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: November 2022-June 2023 Preevaluation: 1 November 2022 Postevaluation: June 2023 Follow up evaluation Januar 2024
- Therapy Group B: Therapy Group B Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  Monthly psychiatric treatment twice a week IPT and MCT, 60 minutes every session
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: November 2022-June 2023 Preevaluation: 1 November 2022 Postevaluation: June 2023 Follow up evaluation Januar 2024
  1. olanzapine 10 mg
  2. clozapine 350 mg, alprazolami 0, 5mg
- Therapy Group C: Therapy Group C Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  Monthly psychiatric treatment twice a week IPT and MCT, 60 minutes every session
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: November 2022-June 2023 Preevaluation: 1 November 2022 Postevaluation: June 2023 Follow up evaluation Januar 2024
  1. Clozapine 250 mg, aripiprazole 10 mg, alprazolam 0.5 mg
  2. olanzapine 30 mg, amisulpride 400 mg
  3. perphenazine 16 mg, olanzapine 10 mg, amitriptyline 40 mg
  4. perphenazine 12 mg, amitriptyline 30 mg, olanzapine 15 mg
  5. aripripazole depot 400 mg, zypahera 405 mg depot
  6. 2 aripripazole depot 400mg (800)
  7. clozapine 400 mg, valproide natrio 1000 mg, stelazine 15 mg
  8. clozapine 300 mg, risperidone 6 mg
- Therapy Group D: Therapy Group D Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  Monthly psychiatric treatment twice a week IPT and MCT, 60 minutes every session
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: Januar 2023-August 2023 Preevaluation: December 2022 Postevaluation: August 2023 Evaluation in follow up: March 2024
  1. clozapine 300mg
  2. clozapine 700mg
  3. clozapine 800mg
  4. clozapine 400 mg, perphenazine 8 mg, 20mg amitriptyline, amisulpride 600 mg
  5. acenapine 20mg, clozapine 200mg
  6. chlopromazine 500 mg, aloperidine 10 mg
  7. chloropromazine 400 mg, 20 mg stelazine (triphioriopromazine)
  8. Risperdal Consta 2, 50 mg, chlopromazine 200 mg
- Therapy Group E: Therapy Group E Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  Monthly psychiatric treatment twice a week IPT and MCT, 60 minutes every session
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: Januar 2023-August 2023 Preevaluation: December 2022 Postevaluation: August 2023 Evaluation in follow up: March 2024
  1. Risperdal consta 50 mg, clozapine 300 mg
  2. paliperidone 9 mg, Chloropromazine 200 mg
  3. aripripazole 60 mg
- Therapy Group F: Therapy Group F Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  Monthly psychiatric treatment twice a week IPT and MCT, 60 minutes every session
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: Januar 2023-August 2023 Preevaluation: December 2022 Postevaluation: August 2023 Evaluation in follow up: March 2024
  1. amisulpride 1200 mg
  2. aloperidine 30 mg, clozapine 200 mg
  3. amisulpride 800 mg
- Therapy Group G: Therapy Group G Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented Monthly psychiatric treatment twice a week IPT and MCT, 60 minutes every session
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: Januar 2023-August 2023 Preevaluation: December 2022 Postevaluation: August 2023 Evaluation in follow up: March 2024
  1. Risperidone 12 mg, akineton 4 mg
  2. clozapine 350 mg
  3. clozapine 400 mg
- Therapy Group H: Therapy Group H Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  Monthly psychiatric treatment twice a week IPT and MCT, 60 minutes every session
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: Januar 2023-August 2023 Preevaluation: December 2022 Postevaluation: August 2023 Evaluation in follow up: March 2024
  1. clozapine 600 mg
  2. clozapine 600 mg
  3. clozapine 750 mg
Period: T1-T2 (11-2022-6 2023, 1 2023- 8 2023)
Arm/Group | Therapy Group A | Therapy Group B | Therapy Group C | Therapy Group D | Therapy Group E | Therapy Group F | Therapy Group G | Therapy Group H
Started (35) | 5 | 2 | 8 | 8 | 3 | 3 | 3 | 3
Completed (34) | 4 | 2 | 8 | 8 | 3 | 3 | 3 | 3
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Anxiety | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: T1-T3 (11-2022-1-2024; 1 2023-3 2024)
Arm/Group | Therapy Group A | Therapy Group B | Therapy Group C | Therapy Group D | Therapy Group E | Therapy Group F | Therapy Group G | Therapy Group H
Started (35) | 5 | 2 | 8 | 8 | 3 | 3 | 3 | 3
Completed (32) | 4 | 2 | 7 | 7 | 3 | 3 | 3 | 3
Not Completed | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Anxiety | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Therapy Group All Participants (Groups A, B, C, D, E, F, G, H): Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  35 individuals with schizophrenia
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  The Groups A, B, C, D, E, F, G, H have been added to one group. They receive the same intervention.
Arm/Group | Therapy Group All Participants (Groups A, B, C, D, E, F, G, H)
Number analyzed (Participants) | 35
Age, Customized [Mean (Standard Deviation); unit: Years] | 31.02 (4.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 14
Race/Ethnicity, Customized [Number; unit: Greek patients] | 35
Region of Enrollment [Number; unit: participants]
  Greece | 35
WAIS, IQ [Mean (Standard Deviation); unit: Units on a scale] | 86.17 (3.92)

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Functions: Matrics Consensus Cognitive Battery (MCCB), Greek Verbal Test
Description: Greek verbal memory test: (verbal memory semantic condition (average) (minimum 0-maximum 40) (high scores better outcomes) MCCB: (Neuropsychological Assessment Battery) (NAB) (reasoning and problem solving): (minimum 0 maximum 26) (high scores better outcomes) Data is analyzed through SPS 13.
Time Frame: Baseline T1 (preintervention)-follow-up T3 (after 6 months, up to 55 weeks)
Population: All participants in T1, T3. All participants participate in the same therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Therapy Group All Participants: The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: November 2022-March 2024 Preevaluation: 1 November 2022 35 participants
  35 participants
Arm/Group | Therapy Group All Participants
Number analyzed (Participants) | 35
score on a scale
  Verbal memory T1 | 12.09 (1.28)
  Verbal memory T3 | 19.04 (1.70)
  Problem-solving (NAB) T1 | 7.71 (1.80)
  Problem-solving (NAB) T3 | 14.00 (2.12)
Statistical Analysis 1: Comparison: Therapy Group All Participants; Test type: Superiority; p = .00, ANOVA — Bonferroni correction p<.05 F(1.25)=9.17 η=.254 (p<.05)
Statistical Analysis 2: Comparison: Therapy Group All Participants; Test type: Superiority; p = .00, ANOVA — Bonferroni correction p<.05 F(2)=7.30 η=.213 (P<.05)

2. Primary Outcome: Symptoms, PANSS Greek Version
Description: (PANSS) Greek Version Positive symptoms (minimum 8 maximum 49) low scores better outcomes Negative symptoms: (minimum 8 maximum 49) low scores better outcomes General Psychopathology: (minimum 17 maximum 112) low scores better outcomes Total: Sum of positive, negative and general symptoms (minimum 31, maximum 210), low scores better outcomes The total score is used in the statistical analysis
  (PSYRAT)
  Auditory hallucinations (minimum 0 maximum 44) low scores better Delusion (minimum 0 maximum 24) low scores better Data is analyzed with SPSS 13
Time Frame: Baseline T1 (preintervention)-follow-up T3 (after 6 months, up to 55 weeks)
Population: Evaluation of T1, T3. All participants participate in the same therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Therapy Group All Participants: 35 The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: November 2022-March 2024
Arm/Group | Therapy Group All Participants
Number analyzed (Participants) | 35
score on a scale
  PANSStotal T1 | 113.62 (15.49)
  PANSStotal T3 | 70.18 (7.67)
Statistical Analysis 1: Comparison: Therapy Group All Participants; Test type: Superiority; p = .04, ANOVA — F(2)=3.20, η=.106 Bonferroni Correction p<.05

3. Primary Outcome: Functional Outcome
Description: WHO DAS 2.0 WHODAS total: (functional outcome) (minimum 0-maximum 100) low scores better outcomes Data are analyzed with SPSS 13
Time Frame: Baseline T1 (preintervention)-follow-up T3 (after 6 months, up to 55 weeks)
Population: All participants in T1, T3. All participants participate in the same therapy.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Therapy Group All Participants: Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  35 individuals with schizophrenia
Arm/Group | Therapy Group All Participants
Number analyzed (Participants) | 35
score on a scale
  WHODAStotal T1 | 33.47 (24.55)
  WHODAStotal T3 | 30.49 (6.78)
Statistical Analysis 1: Comparison: Therapy Group All Participants; Test type: Superiority; p = .00, ANOVA — F(1,06)=8,11, η2=.231 Bonferroni correction p<.05

4. Primary Outcome: Recovery
Description: RAS-DS scale Total score (sum of the scores) (0-152) high scores are better outcomes
  Data is analyzed through SPSS 13
Time Frame: Baseline T1 (preintervention)-follow-up T3 (after 6 months, up to 55 weeks)
Population: All participants in T1, T3. All participants participate in the same therapy.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Therapy Group All Participants: Intervention:
  Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
Arm/Group | Therapy Group All Participants
Number analyzed (Participants) | 35
score on a scale
  RECOVERY total T1 | 90.62 (16.49)
  RCOVERY total T3 | 125.56 (10.12)
Statistical Analysis 1: Comparison: Therapy Group All Participants; Test type: Superiority; p = .04, ANOVA — F(1,19)=4,30, η2=.137 Bonferroni correction p<0.5

5. Secondary Outcome: Intelligent Quotient
Description: Intelligence, high scores are better Data is analyzed through SPSS 13.
Time Frame: Baseline T1 (preintervention)
Population: Pre-intervention
Measure: Mean (Standard Deviation); unit: score on a scale IQ
Groups:
- Therapy Group All Participants: Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented in patients with schizophrenia
Arm/Group | Therapy Group All Participants
Number analyzed (Participants) | 35
score on a scale IQ | 86.17 (3.92)
Statistical Analysis 1: Comparison: Therapy Group All Participants; Test type: Superiority; p = .00, t-test, 1 sided — t (38.70)

ADVERSE EVENTS:
Time Frame: November 2022-March 2024. Adverse events were evaluated monthly, from Novemeber 2022-March 2024, for every participant.
Description: Our systematic assessment during the study highlighted no risk for serious adverse events, for mortality or for other adverse events
Groups:
- Therapy Group A: Therapy Group A Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  5 individuals with schizophrenia
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: November 2022-June 2023 Preevaluation: October 2022 Postevaluation: June 2023 Follow up evaluation Januar 2024 5 assessed for serious adverse events, 0 affected
- Therapy Group B: Therapy Group B Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  2 individuals with schizophrenia
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: November 2022-June 2023 Preevaluation: October 2022 Postevaluation: June 2023 Follow up evaluation Januar 2024 2 assessed for serious adverse events, 0 affected
- Therapy Group C: Therapy Group C Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  8
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: November 2022-June 2023 Preevaluation: October 2022 Postevaluation: June 2023 Follow up evaluation Januar 2024 8 assessed for serious adverse events, 0 affected
- Therapy Group D: Therapy Group D Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  8
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: Januar 2023-August 2023 Preevaluation: December 2022 Postevaluation: August 2023 Evaluation in follow up: March 2024 8 assessed for serious adverse events, 0 affected
- Therapy Group E: Therapy Group E Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  3
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: Januar 2023-August 2023 Preevaluation: December 2022 Postevaluation: August 2023 Evaluation in follow up: March 2024 3 assessed for serious adverse events, 0 affected
- Therapy Group F: Therapy Group F Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  3
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: Januar 2023-August 2023 Preevaluation: December 2022 Postevaluation: August 2023 Evaluation in follow up: March 2024 3 assessed for serious adverse events, 0 affected
- Therapy Group G: Therapy Group G Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented
  3
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: Januar 2023-August 2023 Preevaluation: December 2022 Postevaluation: August 2023 Evaluation in follow up: March 2024 3 assessed for serious adverse events, 0 affected
- Therapy Group H: Therapy Group H Intervention: Pharmacotherapy in combination with the Integrated Psychological Therapy and Metacognitive Training will be implemented.
  3
  The combination of the Integrated Psychological Therapy and Metacognitive Training in individuals with schizophrenia and treatment resistant schizophrenia: The combination of pharmacotherapy and psychotherapy in individuals with schizophrenia and treatment resistant schizophrenia.
  Therapy period: Januar 2023-August 2023 Preevaluation: December 2022 Postevaluation: August 2023 Evaluation in follow up: March 2024 3 assessed for serious adverse events, 0 affected
Arm/Group | Therapy Group A | Therapy Group B | Therapy Group C | Therapy Group D | Therapy Group E | Therapy Group F | Therapy Group G | Therapy Group H
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2 | 0/8 | 0/8 | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/8 | 0/8 | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/8 | 0/8 | 0/3 | 0/3 | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
No limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT05623228/Prot_SAP_005.pdf
  • Informed Consent Form (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT05623228/ICF_006.pdf